CLINICAL TRIAL: NCT07051551
Title: Evaluation of the Clinical Performance of a Highly Filled Flowable Composite in Class III Cavity Restorations: A Randomized Controlled Clinical Trial
Brief Title: Clinical Performance of a Highly-filled Flowable Composite in Class III Restorations.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Buse Uygunöz, research assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KA-24010
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Dental Caries
Keywords: dental caries; highly filled flowable resin composite; class ııı restorations
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: randomized controlled clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- highly filled flowable resin composite (Experimental): After etching the enamel with 37% phosphoric acid for 30 seconds, the area will be rinsed with water for 20 seconds and gently air-dried. One layer of adhesive (G2 Bond, GC Corp, Tokyo, Japan) will be applied according to the manufacturer's instructions and polymerized for 10 seconds with a LED light curing unit.The injectable composite resin (G-Aenial Universal Injectable) will be placed similarly in 2 mm increments and light-cured.
  Interventions: Device: tooth restoration
- conventional resin composite (Active Comparator): After etching the enamel with 37% phosphoric acid for 30 seconds, the area will be rinsed with water for 20 seconds and gently air-dried. One layer of adhesive (G2 Bond, GC Corp, Tokyo, Japan) will be applied according to the manufacturer's instructions and polymerized for 10 seconds with a LED light curing unit. Conventional composite resin (G-Aenial A'chord) will be placed in increments of no more than 2 mm, each layer light-cured.
  Interventions: Device: tooth restoration

INTERVENTIONS:
Device: tooth restoration — restoration of class ııı cavities
  Arms: conventional resin composite
Device: tooth restoration — restoration of class ııı cavities
  Arms: highly filled flowable resin composite

SUMMARY:
The aim of this study was to evaluate the 12-month clinical performance of a highly filled flowable composite resin in anterior teeth.

The study will include healthy individuals over the age of 18 who apply to the Department of Restorative Dentistry, Faculty of Dentistry, Hacettepe University, for the treatment of Class III lesions in their anterior teeth. After explaining the purpose and procedures of the study, participants will be asked to sign an informed consent form if they agree to participate. Gender, age, and the tooth numbers to be treated will be recorded. A total of 100 maxillary anterior incisor teeth in 50 patients will be treated, ensuring a balanced distribution of treated teeth between the right and left arches.

A split-mouth design will be used, whereby at least two teeth per patient will be included in the study, and each of the two restorative materials will be applied to one tooth. The allocation of restorative material to each tooth will be randomized. Before the procedure, the names of both materials will be written on separate papers, placed into envelopes, and a member of the auxiliary staff will randomly select one envelope during the restoration stage to ensure randomization.

The sample size was calculated using the Sealed Envelope software program (Sealed Envelope Ltd., 2012). It was assumed that 95.0% of the restorations would remain intact over 12 months, with α = 0.05, power = 80%, and an expected 10% difference between groups. Based on these parameters, the required sample size was calculated as 33. Considering the possibility of patient dropout during the study, 50 teeth per group were included.

DETAILED DESCRIPTION:
Objective The objective of this randomized controlled clinical trial is to evaluate the 12-month clinical performance of a highly filled flowable composite resin in the restoration of Class III lesions in anterior teeth.

Study Design and Participants This study will be conducted at the Department of Restorative Dentistry, Faculty of Dentistry, Hacettepe University. A total of 50 healthy adult participants (≥18 years) who present with at least two Class III lesions in their maxillary anterior teeth will be included. The inclusion process will involve verbal and written explanations of the study protocol, and participants who provide written informed consent will be enrolled.

Patient demographic information, including age and gender, as well as the numbers of the teeth to be treated, will be recorded. In total, 100 maxillary anterior teeth (2 per patient) will be restored, with a balanced distribution between the right and left dental arches.

A split-mouth design will be used, where each patient will receive two restorations, each using a different composite resin. The allocation of materials to each tooth will be randomized by sealed-envelope selection to ensure blinding during the restorative procedure.

Sample Size Calculation The required sample size was determined using the Sealed Envelope software (Sealed Envelope Ltd., 2012). Assuming a restoration survival rate of 95% over 12 months, a significance level (α) of 0.05, 80% statistical power, and a 10% expected difference between groups, the minimum required sample size was calculated as 33 restorations. To account for potential dropouts, 50 teeth per group were included.

Group Allocation

Participants' teeth will be randomly assigned to one of the following two groups:

Group 1: Class III lesions restored with G-ænial A'Chord (conventional nanohybrid composite resin, GC).

Group 2: Class III lesions restored with G-ænial Universal Injectable (highly filled flowable composite resin, GC).

Clinical Procedures All restorative procedures will be performed under standardized conditions. Initial cleaning of tooth surfaces will be done using pumice and polishing rubbers. Following rubber dam isolation, cavity preparation will be carried out using round-ended diamond burs under water cooling. Caries removal will be completed using sharp hand instruments and single-use steel burs of appropriate size.

Cavity dimensions (mesio-distal width, inciso-gingival height, and depth) will be measured using a CPI probe and recorded in millimeters. Beveling of enamel margins will not be performed to avoid mechanical retention enhancement.

Enamel will be etched with 37% phosphoric acid for 30 seconds, rinsed for 20 seconds, and gently air-dried. A single layer of G2 Bond (GC Corp., Tokyo, Japan) will be applied according to the manufacturer's instructions and polymerized for 10 seconds using a LED curing unit (GC D-Light Pro).

In Group 1, G-ænial A'Chord will be applied in ≤2 mm increments, each layer cured with LED light.

In Group 2, G-ænial Universal Injectable will be similarly placed in ≤2 mm layers and cured.

Finishing and polishing will be carried out using finishing burs, polishing discs, and rubber instruments.

Inclusion Criteria

Participants must fulfill all of the following criteria to be included in the study:

Be at least 18 years of age.

Have at least two Class III lesions in maxillary anterior teeth.

Lesions must be classified as D2 (involving half the dentin thickness) and must not extend to D3 (three-quarters dentin depth).

Must provide signed informed consent.

Be physically capable of attending all follow-up appointments.

Have no periapical pathology in the involved teeth.

Exclusion Criteria

Participants will be excluded from the study if they meet any of the following conditions:

Presence of severe periodontal disease affecting the tooth planned for restoration.

Absence of an opposing tooth or lack of occlusal function involving the affected tooth.

Subgingival extension of the lesion beyond the cervical margin.

Lesions limited to enamel without dentinal involvement.

Extensive lesions that cannot be restored with a direct restorative technique.

Presence of anterior malocclusion affecting tooth positioning or function.

Individuals with intellectual disabilities that may impair communication or compliance.

Teeth that have been previously restored in the area of interest.

Known allergy to methacrylate monomers or methacrylate-based polymers.

Patients under the age of 18 or over the age of 64.

ELIGIBILITY:
Inclusion Criteria:

Be at least 18 years of age.

Have at least two Class III lesions in maxillary anterior teeth.

Lesions must be classified as D2 (involving half the dentin thickness) and must not extend to D3 (three-quarters dentin depth).

Must provide signed informed consent.

Be physically capable of attending all follow-up appointments.

Have no periapical pathology in the involved teeth.

Exclusion Criteria:

Presence of severe periodontal disease affecting the tooth planned for restoration.

Absence of an opposing tooth or lack of occlusal function involving the affected tooth.

Subgingival extension of the lesion beyond the cervical margin.

Lesions limited to enamel without dentinal involvement.

Extensive lesions that cannot be restored with a direct restorative technique.

Presence of anterior malocclusion affecting tooth positioning or function.

Individuals with intellectual disabilities that may impair communication or compliance.

Teeth that have been previously restored in the area of interest.

Known allergy to methacrylate monomers or methacrylate-based polymers.

Patients under the age of 18 or over the age of 64.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Retention alpha for at least %90 of the restorations | 1 year
  The primary endpoint was the assessment of restoration retention and absence of material fracture, evaluated according to the FDI World Dental Federation clinical criteria. A restoration was considered successful if it received a score of 1 (excellent) or 2 (good) and remained in place without the need for repair or replacement.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided